CLINICAL TRIAL: NCT02292485
Title: Promoting Informed Decisions About Lung Cancer Screening: Lung Cancer Screening Readiness Study
Brief Title: PCORI-CER-1306-03385 Lung Cancer Screening Readiness Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: PA14-0824
Record Dates: First submitted 2014-11-12; First posted 2014-11-17 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Lung Cancer Screening
Keywords: Lung Cancer Screening; LCS; Survey; Questionnaire; Texas Academy of Family Physicians
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Physicians - Texas Academy of Family Physicians: Physicians attending Texas Academy of Family Physicians event asked to fill out an anonymous survey to better understand their readiness to implement lung cancer screening programs in their practice settings. Surveys administered to physicians attending the TAFP education events in Houston, Texas, October 17-19, 2014 and in Dallas, Texas, November 7-9, 2014.
  Interventions: Behavioral: Survey

INTERVENTIONS:
Behavioral: Survey — Physicians complete survey to better understand their readiness to implement lung cancer screening programs in their practice settings. Surveys administered to physicians attending the TAFP education events in Houston, Texas, October 17-19, 2014 and in Dallas, Texas, November 7-9, 2014.
  Other Names: Questionnaire

SUMMARY:
Investigators will administer a brief, anonymous survey at the Texas Academy of Family Physicians (TAFP) annual Primary Care Summit to better understand the readiness of primary care physicians in Texas to implement lung cancer screening programs in their practice settings.

DETAILED DESCRIPTION:
For this project there will be up to 1000 participants. Physicians attending the annual CME event at the Texas Academy of Family Physicians event will be asked to fill out an anonymous survey to better understand their readiness to implement lung cancer screening programs in their practice settings. The surveys will be administered to physicians attending the TAFP education events in Houston, Texas, October 17-19, 2014 and in Dallas, Texas, November 7-9, 2014.

ELIGIBILITY:
Inclusion Criteria:

1. Physicians attending the TAFP education events in Houston, Texas, October 17-19, 2014 and in Dallas, Texas, November 7-9, 2014.

Exclusion Criteria:

N/A

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Physicians attending the TAFP education events in Houston, Texas, October 17-19, 2014 and in Dallas, Texas, November 7-9, 2014.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2014-10-20 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Lung Cancer Screening Program Readiness | 1 day
  Descriptive statistics (eg, rates) used to describe the readiness of primary care physicians to support lung cancer screening programs in their practices.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Volk, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org